CLINICAL TRIAL: NCT01499641
Title: Epidural Steroid Following Discectomy for Herniated Lumbar Disc Reduces Neurological Impairment and Enhances Recovery. A Randomized Study With Two-year Follow-up
Brief Title: Epidural Steroid Following Discectomy for Herniated Disc Reduces Morbidity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northern Orthopaedic Division, Denmark (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: ON-07-011-RAS
Record Dates: First submitted 2011-12-13; First posted 2011-12-26 (Estimated); Last update posted 2014-09-15 (Estimated); Status verified 2014-09

CONDITIONS: Disc Disease
Keywords: discectomy; methylprednisolone; randomized control trial
MeSH Terms: interventions — Methylprednisolone

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Epidural steroid (Active Comparator): 1.0 mL methylprednisolone acetate 40 mg/mL instilled at the decompressed nerve root
  Interventions: Drug: Methylprednisolone
- None epidural steroid (Experimental)
  Interventions: Drug: Methylprednisolone

INTERVENTIONS:
Drug: Methylprednisolone — Epidural methylprednisolone 40 mg or none

SUMMARY:
Focus of this study is evaluation of the outcome, neurologic impairment and safety of epidural steroide following lumbar discectomy for herniated disc disease.

DETAILED DESCRIPTION:
Methylprednisolone might enhance recovery after discectomy for herniated disc disease without apparent side effect.

Convalescence after discectomy for herniated disc disease is dependent on pain and the inflammatory response. In arthroscopic and abdominal surgery steroids reduce the inflammatory response and enhance recovery.

200 patients with herniated disc disease are randomly allocated to receive epidural methylprednisolone 40 mg or none.

ELIGIBILITY:
Inclusion Criteria:

* Patients with primary lumbar herniated disc disease who had received and performed standardized conservative treatment program with intensive exercises
* Patients more than 18 years old

Exclusion Criteria:

* Patients with central or lateral spinal stenosis due to spondylosis or disc degeneration who needed bilateral decompression, laminectomy or fusion
* Patients with cauda equina syndrome who needed acute operative treatment
* Lack of informed consent and inability to read and understand Danish

Ages: 18 Years to 66 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2001-05; Primary Completion 2003-08 (Actual); Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
Symptoms and signs of neurologic impairment and rate of operation during a 2-year follow-up. | 2 years

SECONDARY OUTCOMES:
Hospital stay, back and leg pain and reflex deficit. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Sten Rasmussen, M.D.Sci., Study Chair — Orthopaedic Research Unit, Aalborg University Hospital
Locations (3):
- Denmark (3):
  - Orthopaedic Surgery Research Unit, Aalborg University Hospital, Aalborg
  - Section for Surgical Pathophysiology, Juliane Marie Centre, Rigshospitalet, Copenhagen
  - Department of Orthopaedic Surgery, Vejle and Give Hospital, Vejle